CLINICAL TRIAL: NCT00916149
Title: Cognitive Effects of Treatment of Interictal Discharges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: UCB Young Investigator Research Program (Unknown); National EpiFellows Foundation (Unknown); UCB Pharma (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Beth Ami Leeman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMC111754
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; Cognition; Lamictal; Lamotrigine; Keppra; Levetiracetam
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Levetiracetam (Active Comparator): 12 individuals with epilepsy, 6 of whom experience infrequent focal epileptiform discharges and 6 of whom experience frequent focal discharges. These individuals will be treated with levetiracetam (LEV). They will complete repeated EEG/cognitive testing pre- and post-treatment to assess the effects of LEV on discharge frequency, discharge duration, and cognitive task performance.
  Interventions: Drug: levetiracetam
- Lamotrigine (Active Comparator): 12 individuals with epilepsy, 6 of whom experience infrequent generalized discharges and 6 of whom experience frequent generalized discharges. These individuals will be treated with lamotrigine (LMT). They will complete repeated EEG/cognitive testing pre- and post-treatment to assess the effects of LMT on discharge frequency, discharge duration, and cognitive task performance.
  Interventions: Drug: Lamotrigine
- No treatment (No Intervention): 15 healthy subjects, not receiving anticonvulsant medication, will undergo repeated EEG/cognitive testing as a control.

INTERVENTIONS:
Drug: levetiracetam — The dosage of levetiracetam will begin at 500mg twice per day (bid) for the first 4 days, and increase by 500mg every 5 days thereafter until a goal of 1500mg bid is reached. The subject will then remain on levetiracetam at 1500mg bid for 8 weeks, until the conclusion of the study. Medication will be supplied in 500mg tablets, to be taken orally.
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Lamotrigine — The drug will be supplied in 25, 100 and 150mg tablets, to be taken orally per the titration schedule below:
  The regimen will begin at 25mg once per day for the first two weeks, and increase to 50mg once per day during weeks 3 and 4. In week 5, the subject will take 50mg twice per day (bid). The dosage will increase to 50mg in the morning and 100mg at night during week 6. During week 7 the subject will take 100mg bid. During week 8, the subject will take 100mg in the morning and 150mg at night. At week 9, the subject will reach the target dose of 150mg bid. The subject will then remain on lamotrigine at 150mg bid for 7 weeks, until the conclusion of the study.
  Other Names: Lamictal
  Arms: Lamotrigine

SUMMARY:
The purpose of this study is to determine if levetiracetam (for patients with focal seizures) or lamotrigine (for patients with generalized seizures) reduces the occurrence of interictal discharges. The study investigates the possible correlation between reduction of interictal discharges and improved cognitive performance.

DETAILED DESCRIPTION:
Subjects with seizures will be studied with electroencephalography (EEG) and offered medication for prevention of recurrent seizures. Those with focal seizures will be treated with levetiracetam, and those with generalized seizures will be treated with lamotrigine. Subjects will undergo repeated EEG with concurrent cognitive testing before and after initiation of treatment. The proposed study tests 3 hypotheses: 1. that treatment with levetiracetam will reduce focal interictal epileptiform activity, 2. that treatment with lamotrigine will reduce generalized interictal epileptiform activity, and 3. that the extent of interictal epileptiform activity is inversely associated with performance on neuropsychological batteries and computerized cognitive testing. Repeated cognitive/neuropsychological testing obtained at steady state of the study drug and again after approximately 2 months on the final dosage will serve to evaluate the timecourse of potential cognitive benefits.

ELIGIBILITY:
Inclusion Criteria

* 18-55 years of age
* Normal Intelligence Quotient (IQ ≥ 80) as estimated by the Wechsler Test of Adult Reading (WTAR)
* Able to give consent
* The subject's treating physician is planning to prescribe levetiracetam for focal or lamotrigine for generalized seizure prevention
* Either symptomatic or idiopathic seizures.

Exclusion Criteria:

* Non-native English speaking and/or multilingual
* Frequent seizures, since seizures themselves impair cognitive function and present a confounding variable. Subjects may have no more than one seizure or one cluster of seizures per month, with a cluster of seizures including more than one seizure, but between which the patient returns to baseline. The cluster may occur over no more than two consecutive days in one month.
* Seizure(s) must not have occurred within 3 days of enrollment and testing.
* Those with focal seizures who have evidence of renal disease (creatinine clearance less than 80) will be excluded from participation, as levetiracetam is cleared by the kidney.
* Those with focal seizures who have neutrophil counts <1000/microliter will be excluded from participation, as levetiracetam may lower white blood cell counts.
* Those with focal seizures and irritability or mood swings will not be eligible for participation, as levetiracetam may exacerbate these symptoms. This will be determined by self-report, information obtained from the referring physician and medical record.
* Those with generalized seizures who have moderate to severe liver dysfunction (Child-Pugh Grades B and C) will be excluded from participation, as lamotrigine is cleared by the liver and the proposed dosing may not be tolerable in this population. This will be determined by self-report, information obtained from the referring physician, a comprehensive metabolic panel (routinely obtained in new-onset seizures) and the medical record.
* Subjects who are pregnant will not be eligible to take part in the study, as levetiracetam and lamotrigine are classified as Pregnancy Category C drugs and may pose risk to the fetus. Women of childbearing potential will have a urine pregnancy test prior to participation in the study. The urine pregnancy test will be repeated at the final study visit. Subjects with epilepsy who are of childbearing potential must use acceptable methods of birth control during the study, to be continued until one month after discontinuation of the study drug. If a subject does become pregnant during this time period, she must notify the investigators.
* Women who are breastfeeding may not participate in this study. Levetiracetam and lamotrigine may pass into the breastmilk of nursing mothers, posing a risk to the baby.
* Hypersensitivity to lamotrigine, levetiracetam or any components of these products

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Hoch, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Aarts JH, Binnie CD, Smit AM, Wilkins AJ. Selective cognitive impairment during focal and generalized epileptiform EEG activity. Brain. 1984 Mar;107 ( Pt 1):293-308. doi: 10.1093/brain/107.1.293. PMID 6421454
- [Background] Browne TR, Penry JK, Proter RJ, Dreifuss FE. Responsiveness before, during, and after spike-wave paroxysms. Neurology. 1974 Jul;24(7):659-65. doi: 10.1212/wnl.24.7.659. No abstract available. PMID 4858089
- [Background] Dodrill CB, Wilkus RJ. Relationships between intelligence and electroencephalographic epileptiform activity in adult epileptics. Neurology. 1976 Jun;26(6 PT 1):525-31. doi: 10.1212/wnl.26.6.525. PMID 819859
- [Background] Gallagher MJ, Eisenman LN, Brown KM, Erbayat-Altay E, Hecimovic H, Fessler AJ, Attarian HP, Gilliam FG. Levetiracetam reduces spike-wave density and duration during continuous EEG monitoring in patients with idiopathic generalized epilepsy. Epilepsia. 2004 Jan;45(1):90-1. doi: 10.1111/j.0013-9580.2004.39503.x. No abstract available. PMID 14692914
- [Background] Goode DJ, Penry JK, Dreifuss FE. Effects of paroxysmal spike-wave on continuous visual-motor performance. Epilepsia. 1970 Sep;11(3):241-54. doi: 10.1111/j.1528-1157.1970.tb03888.x. No abstract available. PMID 5276416
- [Background] Hermann BP, Seidenberg M, Schoenfeld J, Peterson J, Leveroni C, Wyler AR. Empirical techniques for determining the reliability, magnitude, and pattern of neuropsychological change after epilepsy surgery. Epilepsia. 1996 Oct;37(10):942-50. doi: 10.1111/j.1528-1157.1996.tb00531.x. PMID 8822692
- [Background] HOVEY HB, KOOI KA. Transient disturbances of thought processes and epilepsy. AMA Arch Neurol Psychiatry. 1955 Sep;74(3):287-91. doi: 10.1001/archneurpsyc.1955.02330150053007. No abstract available. PMID 13248285
- [Background] Kasteleijn-Nolst Trenite DG, Riemersma JB, Binnie CD, Smit AM, Meinardi H. The influence of subclinical epileptiform EEG discharges on driving behaviour. Electroencephalogr Clin Neurophysiol. 1987 Aug;67(2):167-70. doi: 10.1016/0013-4694(87)90040-x. PMID 2439294
- [Background] KOOI KA, HOVEY HB. Alterations in mental function and paroxysmal cerebral activity. AMA Arch Neurol Psychiatry. 1957 Sep;78(3):264-71. No abstract available. PMID 13457501
- [Background] Lee S, Sziklas V, Andermann F, Farnham S, Risse G, Gustafson M, Gates J, Penovich P, Al-Asmi A, Dubeau F, Jones-Gotman M. The effects of adjunctive topiramate on cognitive function in patients with epilepsy. Epilepsia. 2003 Mar;44(3):339-47. doi: 10.1046/j.1528-1157.2003.27402.x. PMID 12614389
- [Background] Lutz MT, Helmstaedter C. EpiTrack: tracking cognitive side effects of medication on attention and executive functions in patients with epilepsy. Epilepsy Behav. 2005 Dec;7(4):708-14. doi: 10.1016/j.yebeh.2005.08.015. Epub 2005 Nov 2. PMID 16266826
- [Background] Meador KJ, Loring DW, Vahle VJ, Ray PG, Werz MA, Fessler AJ, Ogrocki P, Schoenberg MR, Miller JM, Kustra RP. Cognitive and behavioral effects of lamotrigine and topiramate in healthy volunteers. Neurology. 2005 Jun 28;64(12):2108-14. doi: 10.1212/01.WNL.0000165994.46777.BE. PMID 15985582
- [Background] The Psychological Corporation. Wechsler Test of Adult Reading. 2001, San Antonio, TX: Harcourt Assessment
- [Background] Schwab RS. Research Publications. Reaction time in petit mal epilepsy. Association for Research in Nervous and Mental Disease 1947; 26:339-341.
- [Background] Selldén U. Psychotechnical performance related to paroxysmal discharges in EEG. Clinical Electroencephalography 1971; 2:18-27.
- [Background] Shewmon DA, Erwin RJ. The effect of focal interictal spikes on perception and reaction time. I. General considerations. Electroencephalogr Clin Neurophysiol. 1988 Apr;69(4):319-37. doi: 10.1016/0013-4694(88)90004-1. PMID 2450731
- [Background] Shewmon DA, Erwin RJ. The effect of focal interictal spikes on perception and reaction time. II. Neuroanatomic specificity. Electroencephalogr Clin Neurophysiol. 1988 Apr;69(4):338-52. doi: 10.1016/0013-4694(88)90005-3. PMID 2450732
- [Background] Synder, P.J. Epilepsy. In Snyder, P.J. & Nussbaum, P.D, Clinical neuropsychology: a pocket handbook for assessment. 1998, Washington DC: American Psychological Association.
- [Background] Stodieck S, Steinhoff BJ, Kolmsee S, van Rijckevorsel K. Effect of levetiracetam in patients with epilepsy and interictal epileptiform discharges. Seizure. 2001 Dec;10(8):583-7. doi: 10.1053/seiz.2001.0582. PMID 11792161
- [Background] Stroup E, Langfitt J, Berg M, McDermott M, Pilcher W, Como P. Predicting verbal memory decline following anterior temporal lobectomy (ATL). Neurology. 2003 Apr 22;60(8):1266-73. doi: 10.1212/01.wnl.0000058765.33878.0d. PMID 12707428
- [Background] TIZARD B, MARGERISON JH. THE RELATIONSHIP BETWEEN GENERALIZED PAROXYSMAL E.E.G. DISCHARGES AND VARIOUS TEST SITUATIONS IN TWO EPILEPTIC PATIENTS. J Neurol Neurosurg Psychiatry. 1963 Aug;26(4):308-13. doi: 10.1136/jnnp.26.4.308. No abstract available. PMID 14043044
- [Background] Tizard B, Margerison JH. Psychological functions during wave-spike discharge. British Journal of Social and Clinical Psychology 1963b; 3:6-15.
- [Background] Tromp SC, Weber JW, Aldenkamp AP, Arends J, vander Linden I, Diepman L. Relative influence of epileptic seizures and of epilepsy syndrome on cognitive function. J Child Neurol. 2003 Jun;18(6):407-12. doi: 10.1177/08830738030180060501. PMID 12886976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 subjects enrolled in the Lamotrigine arm. They underwent study procedures, including EEG. The study aim was to compare subjects with and without frequent discharges on EEG. None of these subjects had frequent discharges, and no additional subjects could be recruited. Hence, planned comparisons could not be made and the data were not analyzed.
Groups:
- No Treatment: Healthy subjects, not receiving anticonvulsant medication, will undergo repeated EEG/cognitive testing as a control.
- Levetiracetam: Individuals with epilepsy who will be treated with levetiracetam (LEV). They will complete repeated EEG/cognitive testing pre- and post-treatment to assess the effects of LEV on discharge frequency, discharge duration, and cognitive task performance.
- Lamotrigine: Individuals with primary generalized epilepsy, who will be treated with lamotrigine (LMT). They will complete repeated EEG/cognitive testing pre- and post-treatment to assess the effects of LMT on discharge frequency, discharge duration, and cognitive task performance.
Period: Overall Study
Arm/Group | No Treatment | Levetiracetam | Lamotrigine
Started | 16 | 10 | 5
Completed | 12 | 8 | 5
Not Completed | 4 | 2 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Unable to place scalp EEG leads | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 controls enrolled in "no treatment"; 1 subject did not perform tests due to vision loss and difficulty placing EEG leads. Hence, there are 15 subjects in the "no treatment" arm.
  We were unable to recruit any subjects with generalized epilepsy and frequent discharges, hence we did not complete the analysis of this arm as planned.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment | Levetiracetam | Lamotrigine | Total
Number analyzed (Participants) | 15 | 10 | 5 | 30
Age, Continuous [Mean (Full Range); unit: years] | 31.4 [18 to 43] | 35.8 [22 to 50] | 31.4 [18 to 43] | 35.3 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 4 | 18
  Male | 6 | 5 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 4
  White | 11 | 9 | 5 | 25
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Focal Interictal Discharges (IEDs) Per Hour, Pre to Post Treatment
Description: This descriptive analysis examined the change in interictal discharge rates pre to post-treatment with levetiracetam in subjects with epilepsy and with no treatment in healthy controls.
Time Frame: 1 and 11 weeks
Population: In a preliminary analysis, data from 11 healthy controls and 6 subjects with partial-onset epilepsy were evaluated.
Measure: Mean (Standard Deviation); unit: IEDs/hour
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
IEDs/hour | -28.8 (71.8) | .54 (1.44)
Statistical Analysis 1: Comparison: No Treatment vs Levetiracetam; Change in frequency of IEDs/per hour was assessed for each group (levetiracetam and no treatment); Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test — For each group (levetiracetam and no treatment), the change in IEDs/hour from pre to post-intervention: p >0.05. The a priori threshold for statistical significance was p=0.05

2. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: CVLT Trial 1 Learning Score
Description: Change in California Verbal Learning Test (CVLT) Trial 1 learning score (range 0-16; higher score indicates better memory)
Time Frame: 1 and 11 weeks
Population: Not all subjects completed each neuropsychological test (e.g., lack of time, fatigue, computer issues); hence, the number analyzed may differ across measures.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
scores on a scale | 2.45 (1.29) | 2.5 (2.88)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the CVLT Trial 1 Learning Score from pre to post time points in the no treatment group; Test type: Other; p = 0.005, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the CVLT Trial 1 Learning Score from pre to post time points in the levetiracetam group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

3. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: CVLT Total Learning
Description: Change in California Verbal Learning Test (CVLT) Total Learning Score (the total learning score is summed across 5 learning trials, range 0-80). Higher scores indicate better memory. Scores on the CVLT reflect the number of words recalled.
Time Frame: 1 and 11 weeks
Population: Not all subjects completed each neuropsychological test (e.g., lack of time, fatigue, computer issues); hence, the number analyzed may differ across outcome measures.
Measure: Mean (Standard Deviation); unit: number recalled
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
number recalled | 8.09 (8.79) | 5.5 (6.78)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the CVLT Total Learning Score from pre to post time points in the no treatment group; Test type: Other; p = 0.016, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the CVLT Total Learning Score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

4. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: CVLT Short Delay
Description: Change in California Verbal Learning Test (CVLT) Short Delay Recall Score (the score ranges from 0-16, reflecting the number of words recalled)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number recalled
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 5
number recalled | 1.27 (2.65) | -0.4 (2.07)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the CVLT Short Delay score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the CVLT Short Delay score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

5. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: CVLT Long Delay
Description: Change in California Verbal Learning Test (CVLT) Long Delay Recall score (the score ranges from 0-16, reflecting the number of words recalled)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number recalled
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
number recalled | 1.55 (3.21) | 2.67 (2.16)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the CVLT Long Delay score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the CVLT Long Delay score from pre to post time points in the levetiracetam treatment group; Test type: Other; p = 0.045, Wilcoxon Signed Ranks Test

6. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: BVMT-R Learning
Description: Change in Brief Visuospatial Memory Test-Revised (BVMT-R) Learning score (the score ranges from 0-6, reflecting the number of shapes recalled on the initial learning trial)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number recalled
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
number recalled | .45 (1.92) | .33 (1.63)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the BVMT-R Learning score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the BVMT-R Learning score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

7. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: BVMT-R Total Learning
Description: Change in Brief Visuospatial Memory Test-Revised (BVMT-R) Total Learning score (the score is summed across 3 learning trials, score range 0-18, reflecting the total number of shapes recalled)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number recalled
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
number recalled | 1.09 (3.05) | .17 (2.93)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the BVMT-R Total Learning score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the BVMT-R Total Learning score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

8. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: BVMT-R Delayed Recall
Description: Change in Brief Visuospatial Memory Test-Revised (BVMT-R) Delayed Recall score (the score ranges from 0-6, reflecting the number of shapes recalled after a 25 minute delay)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number recalled
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
number recalled | .36 (.81) | .33 (.52)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the BVMT-R Delayed Recall score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the BVMT-R Delayed Recall score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

9. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: QOLIE
Description: Change in Quality of Life Inventory in Epilepsy-89 score (QOLIE; score ranges from 0-100; higher scores reflect better quality of life)
Time Frame: 1 and 11 weeks
Population: Not all subjects completed each neuropsychological test (e.g., lack of time, fatigue, computer issues); hence, the number analyzed may differ across outcome measures. The QOLIE is specific to epilepsy and was only administered in that subject group.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 0 | 6
scores on a scale |  | 19.6 (27.8)
Statistical Analysis 1: Comparison: Levetiracetam; This analysis assessed the change in the QOLIE score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

10. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: LNS
Description: Change in Letter-Number Sequencing score (LNS; score ranges from 0-21; higher scores indicate better performance). The score reflects the number of items that the subject can correctly recall and place in proper alphabetical and numerical sequence.
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
scores on a scale | .18 (1.66) | -0.5 (1.98)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Letter Number Sequencing score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Letter Number Sequencing score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

11. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Spatial Span
Description: Change in Spatial Span score (score ranges from 0-32; higher scores indicate better performance). Scores indicate the number of spatial sequences correctly recalled, forwards and backwards.
Time Frame: 1 and 11 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number recalled
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
number recalled | .36 (3.08) | -1.67 (1.51)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Spatial Span score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Spatial Span score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

12. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Digit Span
Description: Change in Digit Span score (score ranges from 0-30; higher scores indicate better performance). Scores indicate the number of digit sequences correctly recalled, forwards and backwards.
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number recalled
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
number recalled | .73 (4) | -.33 (2.81)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Digit Span score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Digit Span score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

13. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Verbal Fluency
Description: Change in Verbal Fluency score (Score range: lowest score = 0, with no upper limit, reflecting total number of words generated. Higher scores indicate better performance.)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
scores on a scale | -1.55 (11.26) | -.83 (12.95)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Verbal Fluency score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Verbal Fluency score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

14. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Stroop
Description: Change in Stroop score (The score is the time for completion in seconds; less time reflects better performance.)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 9 | 6
seconds | .98 (12.15) | -7.3 (14.19)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in Stroop performance from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in Stroop performance from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

15. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Design Fluency
Description: Change in Design Fluency score (Score range: lowest score = 0; there is no upper limit. A higher score reflects more designs generated, hence better performance.)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 10 | 6
scores on a scale | 2.8 (4.52) | .83 (3.97)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Design Fluency score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Design Fluency score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

16. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Trails Test
Description: Change in Trails Test score (The score is the time for completion in seconds. A lower score reflects better performance.)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 10 | 6
seconds | -9.51 (18.73) | 11.29 (16.4)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in performance on the Trails Test from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in performance on the Trails Test from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

17. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Grooved Pegboard
Description: Change in Grooved Pegboard Score (The score is the time for completion. A lower score reflects better performance.)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 9 | 6
seconds | -4.73 (18.9) | -4.36 (23.94)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in performance on the Grooved Pegboard task from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in performance on the Grooved Pegboard task from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

18. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Digit Symbol
Description: Change in Digit Symbol Score (The score is the number of items completed. A higher score reflects better performance.)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 10 | 6
scores on a scale | 3.2 (2.78) | 1.5 (3.02)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Digit Symbol score from pre to post time points in the no treatment group; Test type: Other; p = 0.014, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Digit Symbol score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

19. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: CPT Accuracy
Description: Change in Continuous Performance Test Score - Accuracy (CPT; score ranges from 0-100% correct)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
percentage of correct responses | -0.01 (0.03) | .01 (.03)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the CPT Accuracy score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the CPT Accuracy score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

20. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: CPT Reaction Time (CPT RT)
Description: Change in Continuous Performance Test Score - Reaction Time, measured in seconds (CPT RT; less time reflects better performance)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
seconds | 1.04 (110.54) | -11.33 (52.77)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the CPT reaction time from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the CPT reaction time from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

21. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Choice Accuracy
Description: Change in Choice Accuracy Score (indicate if red or blue stimulus; accuracy 0-100%)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 4 | 1
percentage of correct responses | .02 (.01) | .1 (NA) — one one data point obtained, hence no standard deviation can be calculated
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Choice Accuracy score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

22. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Choice Reaction Time
Description: Change in Choice Reaction Time Score, with reaction time measured in seconds (indicate if red or blue stimulus; lower reaction time suggests better performance)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
seconds | 34.96 (51.16) | .45 (95.62)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Choice Reaction Time score from pre to post time points in the no treatment group; Test type: Other; p = 0.05, Wilcoxon Signed Ranks Test

23. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Verbal Working Memory Accuracy
Description: Change in Verbal Working Memory Accuracy Score (range 0-100%)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
percentage of correct responses | 0 (.02) | -.02 (.02)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Verbal Working Memory Accuracy score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Verbal Working Memory Accuracy score from pre to post time points in the levetiracetam treatment group; Test type: Other; p = 0.039, Wilcoxon Signed Ranks Test

24. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Verbal Working Memory Reaction Time
Description: Change in Verbal Working Memory Reaction Time Score, with reaction time measured in seconds (indicates processing speed)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
seconds | -54.76 (112.04) | -9.36 (155.16)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Verbal Working Memory Reaction Time from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Verbal Working Memory Reaction Time from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

25. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Non-verbal Working Memory Accuracy
Description: Change in Non-verbal Working Memory Accuracy Score (accuracy ranges from 0-100%)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
percentage of correct responses | -.01 (.03) | 0 (.02)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Non-verbal Working Memory Accuracy score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Non-verbal Working Memory Accuracy score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

26. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Non-verbal Working Memory Reaction Time
Description: Change in Non-verbal Working Memory Reaction Time Score (indicates processing speed, with reaction time measured in seconds)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
seconds | -31.99 (85.18) | -25.54 (131.96)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Non-verbal Working Memory Reaction Time from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Non-verbal Working Memory Reaction Time from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

27. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Verbal Recognition Accuracy
Description: Change in Verbal Recognition Accuracy Score (accuracy ranges from 0-100%)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 5
percentage of correct responses | .02 (.11) | .14 (.27)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Verbal Recognition Accuracy score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Verbal Recognition Accuracy score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

28. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Verbal Recognition Reaction Time
Description: Change in Verbal Recognition Reaction Time Score (indicates processing speed, with reaction time measured in seconds)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 5
seconds | 2.98 (93.5) | -6.1 (98.44)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Verbal Recognition Reaction Time from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Verbal Recognition Reaction Time from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

29. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Facial Recognition Accuracy
Description: Change in Facial Recognition Accuracy Score (accuracy ranges from 0-100%)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 5
percentage of correct responses | .01 (.17) | .03 (.06)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Facial Recognition Accuracy score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Facial Recognition Accuracy score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

30. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Facial Recognition Reaction Time
Description: Change in Facial Recognition Reaction Time Score (indicates processing speed, with reaction time measured in seconds)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 5
seconds | -66.76 (168.66) | .61 (50.91)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the Facial Recognition Reaction Time from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the Facial Recognition Reaction Time from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

31. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: NDDIE
Description: Change in Neurological Disorders Depression Inventory for Epilepsy (NDDIE) score (scores range from 0-24; higher scores indicate greater depressive symptoms)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
scores on a scale | 0.18 (2.52) | 1.5 (4.28)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the NDDIE score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the NDDIE score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

32. Secondary Outcome: Performance on Neuropsychological Batteries and Computerized Cognitive Testing: Adverse Events Profile (AEP)
Description: Change in Adverse Events Profile score (scores range from 19-76; higher scores indicate greater side effects)
Time Frame: 1 and 11 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No Treatment | Levetiracetam
Number analyzed (Participants) | 11 | 6
scores on a scale | -1.27 (6.75) | 1 (9.01)
Statistical Analysis 1: Comparison: No Treatment; This analysis assessed the change in the AEP score from pre to post time points in the no treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: Levetiracetam; This analysis assessed the change in the AEP score from pre to post time points in the levetiracetam treatment group; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

ADVERSE EVENTS:
Groups:
- Levetiracetam: 8 individuals with focal-onset epilepsy. These individuals 12will be treated with levetiracetam (LEV). They will complete repeated EEG/cognitive testing pre- and post-treatment to assess the effects of LEV on discharge frequency, discharge duration, and cognitive task performance.
- Lamotrigine: 5 individuals with generalized epilepsy. These individuals will be treated with lamotrigine (LMT). They will complete repeated EEG/cognitive testing pre- and post-treatment to assess the effects of LMT on discharge frequency, discharge duration, and cognitive task performance.
- No Treatment: 12 healthy subjects, not receiving anticonvulsant medication, will undergo repeated EEG/cognitive testing as a control.
Arm/Group | Levetiracetam | Lamotrigine | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/12
Other Adverse Events (participants affected / at risk) | 0/8 | 1/5 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=8) | Lamotrigine (N=5) | No Treatment (N=12)
Weight loss (General disorders) | 0 (0) | 1 (1) | 0 (0)
Frustration during cognitive testing (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No